CLINICAL TRIAL: NCT03950934
Title: Classification and Prediction of Difficult Videolaryngoscopic Intubation in Patients Undergoing Oral and Maxillofacial or Ear, Nose and Throat Surgery
Brief Title: Videolaryngoscopic Intubation and Difficult Airway Classification
Acronym: VIDiAC
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV5856
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Oral Surgery; Maxillofacial Surgery
Keywords: Anesthesia; Airway Management; Intubation; Bronchoscopes; Risk Assessment; Surgery
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention, observational study, perioperative survey — no intervention

SUMMARY:
Primary aim of this study is to identify independent factors associated with difficult videolaryngoscopic intubation in patients undergoing oral and maxillofacial (OMF) or ear, nose and throat (ENT) surgery. Furthermore, this study intends to assess the diagnostic value of preoperative flexible nasal videoendoscopy to predict difficult videolaryngoscopic intubation in these patients.

DETAILED DESCRIPTION:
Difficult endotracheal intubation is a major reason for anesthesia related adverse events. Videolaryngoscopy has become an important part of the anesthesiological standard of care for difficult airway management in the past decades. Still, medical preconditions, as well as procedural and technical factors related with difficult videolaryngoscopy have not been systematically investigated, and a standardized comprehensive classification system for the severity of videolaryngoscopic intubation has yet to be specified. The primary objective of this study is to identify independent factors associated with difficult videolaryngoscopic intubation in patients undergoing ENT or OMF surgery.

Patients with conditions of the ENT and OMF spectrum have a predisposition for difficult airway management and are at high risk for adverse events during endotracheal intubation. However, current recommendations for preoperative screening for difficult intubation rarely consider space consuming lesions of the laryngopharyngeal region. Comprehensive data identifying the predictive value of preoperative flexible nasal videoendoscopy as a diagnostic measure to anticipate difficult airway management still lack. Thus, secondary aim of this study is to evaluate the diagnostic value and clinical significance of preoperative flexible nasal videoendoscopy to predict difficult videolaryngoscopic intubation in these patients.

Study design:

The investigators conduct a prospective observational study, which includes 400 patients with predicted difficult airway and confirmed indication for flexible nasal videoendoscopy and videolaryngoscopic intubation undergoing ENT or OMF surgery.

Procedural and surgical data as well as medical preconditions will be assessed systematically. The handling anesthetist and two independent observers will be surveyed (structured questionnaire) in order to assess procedural and technical factors related with videolaryngoscopic intubation.

ELIGIBILITY:
Inclusion criteria:

* 18 Years and older
* Patients scheduling for ENT or OMF surgery under general anesthesia with requirement of endotracheal Intubation
* Risk of difficult airway management with confirmed indication for videolaryngoscopic intubation

Exclusion criteria:

* No consent given
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ENT or OMF surgical patients presenting at the Anesthesiology Preassessment Clinic of the University Medical Center Hamburg-Eppendorf for preoperative risk assessment will be checked for eligibility. Repeated inclusions of participators are allowed.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Difficult videolaryngoscopic intubation | 30 minutes after endotracheal intubation
  Questionnaire

SECONDARY OUTCOMES:
Successful first intubation attempt | 30 minutes after endotracheal intubation
  Observation during airway management
Overall success | 30 minutes after endotracheal intubation
  Observation during airway management
Unsuccessful videolaryngoscopy | 30 minutes after endotracheal intubation
  Observation during airway management
Severity of videolaryngoscopic intubation | 30 minutes after endotracheal intubation
  Numeral rating scale
Specific recommendations of the handling anesthetist | 30 minutes after endotracheal intubation
  Questionnaire
Time to successful intubation | 30 minutes after endotracheal intubation
  Observation during airway management
Number of laryngoscopy and intubation attempts | 30 minutes after endotracheal intubation
  Observation during airway management
Lowest oxygen saturation during airway management | 30 minutes after endotracheal intubation
  Observation during airway management
Initial end-tidal carbon dioxide level after successful intubation | 30 minutes after endotracheal intubation
  Observation during airway management
Observed complications during or after induction of general anesthesia | 30 minutes after endotracheal intubation
  Questionnaire
Length of hospital stay | Until hospital discharge up to 3 months after surgery
  Follow-up
All cause in-hospital mortality | Until hospital discharge up to 3 months after surgery
  Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, PD Dr., Principal Investigator — Department of Anesthesiology, University Medical Center Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peters T, Wunsch VA, Siebert H, Kohl V, Breitfeld P, Dankert A, Sasu PB, Dohrmann T, Krause L, Zollner C, Petzoldt M. What Is a Critical Mouth Opening for Macintosh Videolaryngoscopy? Results From a Prospective Observational Study. Anesth Analg. 2025 Oct 30. doi: 10.1213/ANE.0000000000007838. Online ahead of print. PMID 41452604
- [Derived] Wunsch VA, Kohl V, Breitfeld P, Bauer M, Sasu PB, Siebert HK, Dankert A, Stark M, Zollner C, Petzoldt M. Hyperangulated blades or direct epiglottis lifting to optimize glottis visualization in difficult Macintosh videolaryngoscopy: a non-inferiority analysis of a prospective observational study. Front Med (Lausanne). 2023 Nov 30;10:1292056. doi: 10.3389/fmed.2023.1292056. eCollection 2023. PMID 38098848